CLINICAL TRIAL: NCT06474884
Title: A Single-center, Prospective, Cohort Study of the Safety and Efficacy of Single Antiplatelet Therapy After Pipeline Flex with Shield Stent Implantation for Intracranial Aneurysms
Brief Title: The Safety and Efficacy of Single Antiplatelet Therapy After Pipeline Flex with Shield for Intracranial Aneurysms
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: zp930826
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Treatment
Keywords: intracranial aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this study was to evaluate the safety and efficacy of single antiplatelet therapy after Pipeline flex with Shield stent implantation for intracranial aneurysms.

DETAILED DESCRIPTION:
Title：A single-center, prospective, cohort study of the safety and efficacy of Single Antiplatelet therapy after Pipeline flex with Shield stent implantation for intracranial aneurysms.

Purpose：To assess the safety and efficacy of single antiplatelet therapy after Pipeline flex with Shield stent implantation for intracranial aneurysms.

Follow up:The follow-up period was 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unruptured intracranial aneurysms who received the intracranial Pipeline Flex with Shield stent.
2. Vascular conditions:

1) There was no obvious calcification and stenosis of the parent artery. 2) The curvature of the bearing artery is minimal. 3) The parent artery diameter ≥2.5mm

3.According to the committee's assessment, only one Pipeline flex with shield is needed for aneurysm treatment.

4.Before the stent implantation procedure, standard dual antiplatelet therapy should be administered for at least 3 days.

5.Patients with an Modified Rankin Scale(mRS) score of less than 2 on the day of registration.

6.The operation was successful, and immediate postoperative angiography indicated good wall apposition.

Exclusion Criteria:

1. Patients with recurrent aneurysms after interventional treatment or surgical clipping.
2. The patient after stent placement surgery.
3. Aneurysms can have irregular shapes, such as fusiform, blister-type, or dissecting aneurysms.
4. The patient had no history of stroke or aneurysm rupture in the last 3 months.
5. Abnormal platelet function, or platelet count < 100,000 cells/mm³.
6. Known history of allergy to clopidogrel or heparin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this prospective registry includes patients with unruptured intracranial aneurysms suitable for Pipeline Flex with Shield at the operators' discretion.All patients underwent thromboelastography and CYP2C19 genotyping.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete aneurysm occlusion in 6 months | assessed at 6 months after procedure
  The Raymond-Roy occlusion classification (RROC) is an angiographic classification scheme for grading the occlusion of flow diverter treated cerebral aneurysms (class I: complete obliteration, class II: residual neck, class III: residual aneurysm). Higher class represent a worse outcome. The percentage of Success aneurysm occlusion in which class 1 or 2 is achieved on the Raymond-Roy occlusion classification Scale at the 6 months follow-up angiographic assessments will be evaluated.
Hemorrhagic, ischemic events, or neurological deficits occurring within 6 months postoperatively. | assessed at 6 months after procedure
  Ischemic events include intraoperative and postoperative ischemic stroke, transient ischemic attack, stent thrombosis, emergency revascularization, and cerebrovascular death.
  Hemorrhagic events include: symptomatic or asymptomatic intracranial hemorrhagic events (subarachnoid hemorrhage and intracerebral hemorrhage) within 6 months after surgery; or non-intracranial hemorrhagic events (such as skin petechiae, epistaxis, gingival bleeding, gastrointestinal bleeding, genitourinary bleeding, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China